CLINICAL TRIAL: NCT01062191
Title: Flexible Hydrogel Nanoparticle Wound Dressing Allows Greater Joint Range of Motion Compared to Typical Sodium Carboxymethylcellulose Dressing
Brief Title: Altrazeal Range of Motion Study Comparing With Typical Carboxymethyl
Acronym: ROM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: ULURU Inc. (Industry)
Responsible Party: Vincent Gabriel, MD, UTSW Medical Center, Department of Physical Medicine and Rehabilitation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U-C-6U1101
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Burn
Keywords: hydrogel; dressing; burn; joint
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Altrazeal Flexible Hydrogel Nanoparticle Wound Dressing (Experimental): Nanoflex Powder Dressing applied to joint
  Interventions: Device: Altrazeal Flexible Hydrogel Nanoparticle Wound Dressing
- Aquacel AG, typical carboxymethylcellulose dressing (Active Comparator): Sodium CMC dressing control applied to joint
  Interventions: Device: Aquacel AG, typical carboxymethylcellulose dressing

INTERVENTIONS:
Device: Aquacel AG, typical carboxymethylcellulose dressing — 4" X 4", Aquacel silver sheet
  Arms: Aquacel AG, typical carboxymethylcellulose dressing
Device: Altrazeal Flexible Hydrogel Nanoparticle Wound Dressing — Wound dressing
  Arms: Altrazeal Flexible Hydrogel Nanoparticle Wound Dressing

SUMMARY:
The objective of this study is to evaluate the difference in joint range of motion of a new flexible hydrogel nanoparticle wound dressing compared to typical sodium carboxymethylcellulose dressing Aquacel AG for treatment of partial thickness burns.

DETAILED DESCRIPTION:
This is a single center, randomized, single blind therapeutic exploratory study to monitor the range of motion of wounds treated with the new nanoparticle hydrogel dressing compared to the range of motion of wounds treated with existing treatment standard (sodium carboxymethylcellulose dressing) in patients with partial thickness burns. A total of 50 joints will be studied. The patients will be at least 7 years of age.. The Department of Physical Medicine and Rehabilitation at Parkland Hospital and Health System, UT Southwestern, will be asked to enroll enough patients to meet the proposed 50 joint study sites (approximately 3-5 afflicted joints per patient). Children will be included in the patient population if possible. Inclusion criteria for the medical condition will be at least one partial thickness burn that crosses at least one peripheral joint axial to the proximal interphalangeal joints. As a control, the patients will also need to have an unburned contralateral joint without major internal or external joint derangement.

The Primary Investigator will first identify the study site and control site for each patient and take the initial measurements. Trained personnel will apply the bandage to the study site. No secondary bandage will be applied. Typical meticulous wound care and adequate analgesic medical coverage will be provided for the duration of the study. Both the patient and medical staff will be trained on patient use instructions for the dressing. The patients will be monitored for a short time after application of the bandage as part of standard procedure, and the patient is then allowed to go home with instructions for care. Within 2-8 days after application, the dressing will be inspected and range of motion will be measured for both the study site and the control site. Any concomitant treatment (medications, wound care) will be thoroughly documented for the duration of the study. Both dressings are designed to remain on the wound until the bandage falls off, which indicates re-epithelialization of the wound. The dressings should not be removed by the patient or medical staff unless there are signs of infection, deterioration of bandage, or other adverse event. If the bandage falls off, the patient is instructed to immediately call the medical staff.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient is at least 2 years of age;
2. Patient is in general good health;
3. Patient has partial thickness burn that crosses at least one peripheral joint axial to the proximal interphalangeal joints;
4. Patient has one unburned contralateral joint without major internal or external joint derangement to be used as control
5. Patient is willing and able to cooperate with the protocol for 30 days
6. Patient is capable of provided informed consent
7. Patient provides authorization for use and disclosure of protected health information

Exclusion Criteria:

1. Age less than 2 years;
2. Patient has superficial or full thickness burn wounds;
3. Patient has acutely infected wounds;
4. Patient has wounds with surrounding cellulites;
5. Patient has a history of hypersensitivity to any components of either the nanoparticle or sodium hydrocellulose dressing, or any know sensitivities to other hydrogel bandage treatments
6. Patient has a concurrent clinical condition, which in the judgment of the Investigator cold either pose a health risk to the patient while participating in this study, or could potentially influence the outcome of the study;
7. Patient is wearing any type of orthopedic device that may come in contact with the dressing;
8. Patient has history of poor wound healing, history of smoking, history of drug/alcohol abuse, any other skin/immune system condition that would increase likelihood of wound irritation, infection or increase chance of early termination
9. Patient has wound originating from chronic condition
10. Patients with history of any immunodeficiency syndrome or condition
11. Patients who have applied any dressing or medication (OTC or prescription) to the wound (within 48 hours of study? )
12. Patient has participated in a clinical research study within the last 30 days prior to enrollment;
13. Patient is unable to communicate or to cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Range of motion in burned joints with dressing in place as compared to control | Up to 2 weeks

SECONDARY OUTCOMES:
Pain at joint with dressing in place | up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States